CLINICAL TRIAL: NCT05876936
Title: A Prospective, Open Label Study to Assess the 24-hour Intraocular Pressure Pattern Recorded With Triggerfish® in Patients With Open Angle Glaucoma Before and After DSCI
Brief Title: Prospective, Open Label Study to Assess 24hs IOP Recorded With Triggerfish® in Patients With OAG Before and After DSCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left the hospital
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Dr. Kaweh Mansouri, Chef de clinique, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TF-1307
Record Dates: First submitted 2015-04-24; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- contact lens sensor Triggerfish® in patients selected for deep sclerectomy with collagen implant (Other): The contact lens sensor (CLS) SENSIMED Triggerfish® in will be placed on the study eye as selected for deep sclerectomy with collagen implant (DSCI)
  Interventions: Device: contact lens sensor (CLS) SENSIMED Triggerfish®

INTERVENTIONS:
Device: contact lens sensor (CLS) SENSIMED Triggerfish® — contact lens sensor CLS placing and fitting evaluation, 24h recording

SUMMARY:
A prospective, open label study to assess the 24-hour intraocular pressure pattern recorded with SENSIMED Triggerfish® in patients with open angle glaucoma before and after deep sclerectomy with collagen implant

DETAILED DESCRIPTION:
This is a prospective, open label study to assess the 24-hour IOP pattern recorded by SENSIMED Triggerfish® in Open Angle Glaucoma (OAG) patients before and after deep sclerectomy with collagen implant (DSCI).

After having signed and dated the patient informed consent form, patients will undergo an initial ophthalmic examination. The contact lens sensor (CLS) SENSIMED Triggerfish® will be placed on the study eye as selected for DSCI, for a baseline 24-hour IOP pattern recording session (S1), within 7 days preceding the surgical procedure. Patients will remain ambulatory and will be encouraged to follow a schedule as close to his/her usual lifestyle as possible. A patient diary will be distributed for the capture of patient activities during the IOP pattern recording. Upon completion of S1, the contact lens sensor (CLS) SENSIMED Triggerfish® will be removed and a final ophthalmic examination will be conducted. The patient diary will be collected and concomitant medication will be reported. The surgery will be scheduled within 2 days following S1.

Unless contraindicated (e.g. large filtering bleb precluding placement of the contact lens sensor (CLS) SENSIMED Triggerfish®), patients will undergo a second 24-hour contact lens sensor (CLS) SENSIMED Triggerfish® IOP pattern recording session (S2) on the study eye 3 months after the surgical procedure. S2 will start at the same time of day ± 30 min as S1, preferably at a time that allows for sufficient recording of the wake-to-sleep and the sleep-to-wake phases. Prior to S2 and upon completion of thereof, ophthalmic examinations will be conducted and patient diary will be collected. In addition, any specifics regarding the DSCI and medication will be reported. A visual field (VF) assessment will also be performed to evaluate the changes after deep sclerectomy with collagen implant.

Patients will undergo a third 24-hour SENSIMED Triggerfish® IOP pattern recording session (S3) on the study eye 12 months after the surgical procedure. S3 will start at the same time of day ± 30 min as S2, preferably at a time that allows for sufficient recording of the wake-to-sleep and the sleep-to-wake phases. Prior to S3 and upon completion of thereof, ophthalmic examinations will be conducted and patient diary will be collected. In addition, any specifics regarding the deep sclerectomy with collagen implant (DSCI) and medication will be reported. A visual field assessment will also be performed to evaluate the changes after deep sclerectomy with collagen implant (DSCI).This concludes the study for the patients.

Hence, the overall study duration for the patient is limited to 13 months. The study has been planned to recruit at least 40 eligible patients within 11 months from initiation. Hence the overall study duration from the first patient accrued into the study until last patient out equates to about 24 months or less. Allowing for a database lock within 4 weeks of study completion, a preliminary statistical report on the primary efficacy endpoint is foreseen within 2 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Open Angle Glaucoma (OAG)
* Documented glaucomatous Visual Field damage with MD more negative than -2 dB
* Progressing glaucomatous damage justifying a deep sclerectomy with collagen implant (DSCI)
* Aged ≥18 years, of either sex
* Not more than 6 diopters spherical equivalent on the study eye
* Have given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* • History of ocular surgery within the last 3 months on the study eye

  * History of ocular laser treatment on the study eye
  * Corneal or conjunctival abnormality precluding contact lens adaptation on the study eye
  * Severe dry eye syndrome on the study eye
  * Patients with allergy to corneal anesthetic
  * Patients with contraindications for silicone contact lens wear
  * Patients not able to understand the character and individual consequences of the investigation
  * Participation in other clinical research within the last 4 weeks
  * Any other contra-indication listed in the SENSIMED Triggerfish® user manual

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes between the nycthemeral IOP patterns recorded with TF during two 24-hour periods in patients with OAG | Baseline, 3 months and 12 months
  Nycthemeral IOP patterns differences will be evaluated with SENSIMED Triggerfish® recording for two 24hs periods in Open Angle Glaucoma patients comparing from baseline to 3 and 12 months

SECONDARY OUTCOMES:
Changes in diurnal and nocturnal IOP patterns | 3 months and 12 months after deep sclerectomy with collagen implant (DSCI)
  Evaluation of the effect of deep sclerectomy with collagen implant (DSCI) on diurnal and nocturnal IOP patterns
Changes in visual field | 3 months and 12 months after deep sclerectomy with collagen implant (DSCI)
  Determination of changes in visual field
Number of Adverse Events | 3 months and 12 months after deep sclerectomy with collagen implant (DSCI)
  Evaluation of the safety and tolerability evaluation through the number of adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Kaweh Mansouri, Dr MD, Principal Investigator — Univeresity Hospital Geneva
Locations (1):
- University Hospital Geneva, Geneva, Switzerland